CLINICAL TRIAL: NCT05210205
Title: Physiological Efficacy and Acceptability of Essential Amino Acid-enhanced and Energy Density-enhanced Combat Ration Products During Multi-stressor Operations
Brief Title: Physiological Response to Protein and Energy-enhanced Food Products During Winter Military Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Norwegian Defense Research Establishment (Unknown); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-19HC
Record Dates: First submitted 2021-12-09; First posted 2022-01-27 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Military Operational Stress Reaction; Malnutrition (Calorie); Weight Loss; Muscle Wasting
MeSH Terms: conditions — Malnutrition; Weight Loss; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EAA-enhanced food products (Experimental): Consume approximately 1500 calories of EAA-enhanced food products plus ad libitum consumption of 3 combat rations each day during training.
  Interventions: Dietary Supplement: EAA
- Energy dense food products (Experimental): Consume approximately 1500 calories of energy dense food products plus ad libitum consumption of 3 combat rations each day during training.
  Interventions: Dietary Supplement: Energy Dense
- Control food products (Active Comparator): Consume approximately 1500 calories of low energy dense food products plus ad libitum consumption of 3 combat rations each day during training.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: EAA — EAA-enhanced protein snack bars
  Arms: EAA-enhanced food products
Dietary Supplement: Energy Dense — Energy dense snack bars (same calories in a smaller volume of food)
  Arms: Energy dense food products
Dietary Supplement: Control — Low energy dense snack bars (same calories in a greater volume of food)
  Arms: Control food products

SUMMARY:
Soldiers commonly lose muscle mass during training and combat operations that produce large energy deficits (i.e., calories burned > calories consumed). Developing new combat ration products that increase energy intake (i.e., energy dense foods) or the amount and quality of protein consumed (i.e., essential amino acid [EAA] content) may prevent muscle breakdown and stimulate muscle repair and muscle maintenance during unavoidable energy deficit. The primary objective of this study is to determine the effects of prototype recovery food products that are energy dense or that provide increased amounts of EAAs (anabolic component of dietary protein) on energy balance, whole-body net protein balance, and indices of physiological status during strenuous winter military training.

DETAILED DESCRIPTION:
Up to 96 Norwegian Soldiers participating in a winter training exercise at the Garrison in Sør-Varanger (GSV) will be enrolled in an approximately 11-day, randomized controlled study. Participants will be randomly assigned at the beginning of the training exercise to groups provided 3 Norwegian Army arctic combat rations and approximately 1500 supplemental calories from food products with increased energy density (EN-DENSE), increased essential amino acids (EAA), or low energy density (CONTROL) each day. Participants will be instructed to consume all of the supplemental food products provided to them and consume the arctic combat rations ad libitum. The effect of consuming EN-DENSE, EAA, or CONTROL food products during strenuous military training on physiological status and recovery will be assessed using dietary analysis, stable isotope methodologies, physical performance measures, gut health analyses, blood sampling, and questionnaires. This design will test the hypothesis that 1) EN-DENSE ration products will attenuate the energy deficit during the training, thereby limiting whole-body protein losses and decrements in physiological status; and 2) the protein-sparing benefit of EAA will limit whole-body protein loss regardless of the energy deficit.

ELIGIBILITY:
Inclusion Criteria:

Male and female Norwegian Soldiers aged 18 years or older participating in the winter training exercise at the Garrison in Sør-Varanger.

Exclusion Criteria:

* Any injury or health condition limiting full participation in the training program.
* Allergies or intolerance to foods used in the study (including but not limited to lactose intolerance/milk allergy) or vegetarian practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-13 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Protein balance | 10 hours
  Use stable isotope methodologies to measure whole-body protein balance
Energy Expenditure | 8 days
  Use stable isotope methodologies to measure energy expenditure during the training exercise.
Energy intake | 8 days
  Use food logs and collect food wrappers to measure energy intake during the training exercise.

SECONDARY OUTCOMES:
Intestinal Permeability | 24 hours
  Use dual sugar test (i.e., sucralose and erythritol) to measure intestinal permeability
Gut microbiome composition | Study days -1 and 9
  Measure changes in fecal bacterial community, diversity, and relative abundance
Vertical jump | Study day 0 and 9
  Measure changes in physical performance as determined by a vertical jump test
Pull Strength Test | Study day 0 and 9
  Measure changes in physical performance as determined by a pull strength test

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Howard, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- Garrison in Sør-Varanger, Kirkenes, Norway

IPD SHARING:
Plan to Share IPD: No